CLINICAL TRIAL: NCT05000489
Title: A Qualitative Study of Contraceptive Choice and Decision-making Among Adolescent and Young Adults Living With Chronic Illness and Medical Complexity: a Focus on Long Acting Reversible Contraception (LARC)
Brief Title: Perceptions of LARC Among AYA With Chronic Illness
Acronym: LARC
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, claudia borzutzky, MD; Program Director, Adolescent Medicine Fellowship, CHLA; Clinical Associate Professor of Pediatrics, Keck School of Medicine, USC, Children's Hospital Los Angeles
Other Study IDs: CHLA-20-00511
Record Dates: First submitted 2021-07-01; First posted 2021-08-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2022-05

CONDITIONS: Chronic Conditions, Multiple
Keywords: long acting reversible contraception; birth control; reproductive health; chronic illness; adolescents; young adults; IUD; LARC
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (13):
- Minors 1: a one-time focus group will be conducted with 16-17 year old patients who have a variety of diagnoses
  Interventions: Other: No intervention being administered
- Minor 2: a one-time focus group will be conducted with 16-17 year old patients who have a variety of diagnoses
  Interventions: Other: No intervention being administered
- Spina Bifida: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Spina Bifida clinic
  Interventions: Other: No intervention being administered
- Pulmonology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the pulmonology clinic
  Interventions: Other: No intervention being administered
- Endocrinology 1: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Endocrinology clinic and have a diagnosis of Type I Diabetes
  Interventions: Other: No intervention being administered
- Endocrinology 2: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Endocrinology clinic and have a diagnosis of Type II Diabetes
  Interventions: Other: No intervention being administered
- Rheumatology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Rheumatology clinic
  Interventions: Other: No intervention being administered
- Gastroenterology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Gastroenterology clinic
  Interventions: Other: No intervention being administered
- Neurology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Neurology clinic
  Interventions: Other: No intervention being administered
- Cardiology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Cardiology clinic
  Interventions: Other: No intervention being administered
- Hematology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Hematology clinic
  Interventions: Other: No intervention being administered
- Nephrology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Nephrology clinic
  Interventions: Other: No intervention being administered
- Oncology: a one-time focus group will be conducted with adult patients (18-21) who are being seen in the Oncology clinic
  Interventions: Other: No intervention being administered

INTERVENTIONS:
Other: No intervention being administered — No intervention will be administered. Each patient will participate in a qualitative focus group discussing their beliefs/attitudes about their reproductive health and birth control

SUMMARY:
The investigators aim to perform a qualitative study exploring attitudes and perceived barriers to Long Acting Reversible Contraception (LARC), both implants and IUDs, among adolescent and young adults (AYA) with chronic illness at CHLA. While the literature examining barriers to LARC uptake is growing, its focus has been on older women and women who are not living with chronic illness. There remains a significant gap in the understanding of:

1. What adolescents and young adults from ethnically diverse, economically underserved communities know about LARCs
2. If and how LARCs fit into their considerations and decision making about contraception choices
3. Perceived barriers to LARC among AYA with chronic medical conditions
4. Information, perceptions, experiences that inform choices that may be unique to AYA living with chronic conditions

Research Objectives

1. Explore the impact of the experience of living with chronic medical conditions on AYA patient attitudes toward and acceptance of LARCs
2. Identify AYA patient concerns and perceptions related to historical coercion and reproductive injustice experienced by minority communities that may reduce acceptance of LARC
3. Explore the relationship between patients' perception of pediatric subspecialty care providers' attitudes regarding sexual health and contraception guidance and patients' attitudes toward and acceptance of LARC
4. Identify factors related to patient's age, family's values, and medical condition, as well as historical events or legacies that may impact preference of implant vs intra-uterine device (IUD), independent of safety/medical contraindications, if choosing a LARC method.
5. Explore other social, cultural or psychological factors that influence perception and represent barriers to LARC access

Hypotheses

1. The impact of chronic illness on AYA sense of bodily autonomy (including self-concept, history of other medical procedures, and concerns around mortality) reduces the attractiveness of LARC methods.
2. The intersectionality of multiple oppressions, including racism, xenophobia, sexism, and historical reproductive coercion and injustice implicitly reduce the attractiveness of LARC methods for AYA patients from minority communities with chronic medical conditions at CHLA.
3. Pediatric subspecialty providers' attitudes about sex, and comfort with providing patient-centered contraception counseling, as perceived by AYA patients, impact AYA patient attitudes towards and acceptance of LARC.
4. Preference of implant vs. IUD is related to patient's age, family values, and type of medical condition, as well as their knowledge of historical events related to contraception in their community, independent of safety/medical contraindications.
5. Additional perceived barriers, including fear or skepticism about LARC conferred by trusted sources of information such as family or social media, reduce the attractiveness and acceptance of LARC by AYA with chronic medical conditions

DETAILED DESCRIPTION:
Long acting reversible contraceptives (LARC), including the subdermal etonogestrel implant, and both the copper and levonogestrel intrauterine devices (IUDs), are recommended as first line birth control methods for adolescents and young adults (AYA) by both the American Academy of Pediatrics and the American College of Obstetricians and Gynecologists. LARC have been noted to be particularly safe for reproductive age AYA with chronic illness, a population that needs and benefits greatly from careful guidance about contraception choice. It is well documented that AYA with chronic illness are often as sexually active as their "healthy" peers, but can face both greater health and psychosocial complications if pregnancy is unplanned, and health risks if their contraceptive method interacts adversely with medication regimes. Additionally, in both pediatric and adult specialty care, despite frequent visits, addressing sexual health issues is often omitted, whether by intent or lack of comfort, or due simply to limited time for visits and the precedence given to the primary disease for which the care is being provided.

While there is growing evidence that AYA females are opting for LARC as their contraceptive method few have explored attitudes towards and acceptance of LARC by AYA with chronic illness. Even less is understood about the impact of AYA perceptions of their subspecialty providers' comfort, knowledge, or ability to counsel around sexual health issues on their contraceptive planning and choices. Additionally, little is known about how medical condition, age or other factors may influence perceptions of type of LARC, i.e., implant vs. IUD, or how they may influence decisions to use either type in this population of AYA. The Contraceptive Choice Study did demonstrate greater interest in and use of the implant over IUDs among younger teens, but there was no qualitative inquiry exploring reasons for this difference by age, that investigators are aware of. Lastly, the recent attention to the reproductive justice framework, including a greater understanding of the historical legacy of institutionalized and structural reproductive coercion of non-Caucasian communities in the United States, sheds light on an even greater knowledge gap regarding the intersectionality of minority ethnicity/race, chronic illness, and attitudes towards LARC among AYA. As research aims to move forward into a model of sexual and reproductive care for transition age youth that is grounded in both reproductive justice and cultural humility, the understanding of this intersection becomes critical.

Los Angeles County is one of the most demographically, culturally, and linguistically diverse urban metropolitan areas in the world. The patient populations served by Children's Hospital Los Angeles (CHLA) mirror this diversity. In 2018, CHLA provided care to 133,325 unique patients. Currently, 11,970 adolescents and young adults between 16-21 years of age are receiving care for chronic illness or disability. Over half (52%) are female. Many of CHLA's patients come from immigrant families with limited education and ability to communicate in English. Nearly 60% of CHLA's patients identify as Latinx/Hispanic, and while many adolescent and young adult patients' parents/caretakers are monolingual Spanish speaking, most patients are bilingual in Spanish and English. Over three-quarters (76%) of CHLA's patients rely on Medicaid and Title V benefits for their care. Ranked 5th best pediatric tertiary care institution in the U.S., CHLA is the only pediatric institution among the nation's top 10 to serve as a safety net provider. In fact, CHLA provides care to over a third of Los Angeles county's children with special healthcare needs eligible for Title V benefits. Investigators anticipate that the patients participating in this study will reflect this same ethnic/racial, socio-economic, and cultural diversity.

CHLA's AYA patients are affected by a group of conditions that reflect diversity in their degree of visibility and physical disability, chronicity vs intermittency, number of organ systems involved, and types of treatments. The study team's interest is therefore to also explore differences in attitudes, behavior and perceptions toward LARC that may relate to the nature of their particular condition and treatment regimen.

The CHLA Division of Adolescent and Young Adult Medicine serves as the primary sexual/reproductive health referral point for CHLA's AYA patients with chronic illness; it has offered placement of the etonogestrel implant since shortly after it was introduced into the U.S. market by Organon, and has offered IUD placements since spring of 2017. However, uptake of LARC among CHLA AYA patients is low. Since 2013, approximately 200 LARCs have been placed; approximately 30 were placed in 2019.

The study team's aim is to perform a qualitative study exploring attitudes and perceived barriers to LARC, both implants and IUDs, among AYA with chronic illness at CHLA. While the literature examining barriers to LARC uptake is growing, its focus has been on older women and women who are not living with chronic illness. There remains a significant gap in the understanding of:

1. What adolescents and young adults from ethnically diverse, economically underserved communities know about LARCs
2. If and how LARCs fit into their considerations and decision making about contraception choices
3. Perceived barriers to LARC among AYA with chronic medical conditions
4. Information, perceptions, experiences that inform choices that may be unique to AYA living with chronic conditions

This observational study will employ qualitative methods targeting adolescent and young adult (AYA) females 16-21 years of age living with chronic illness or disability. A key research question underlying these themes will be to explore the extent to which their experiences living with chronic illness and their engagement in ongoing medical management has an impact on their contraception decision making and perception of LARC as a viable option.

Approximately 90-110 sexually active and non-sexually active young women or transmale identified (have the potential for pregnancy) 18-21 years of age who are receiving ongoing healthcare from subspecialty teams at Children's Hospital Los Angeles will be recruited to participate in a one-time focus group session, with the focus group being comprised of 5-10 individuals each. There is expected to be 11 adult aged focus groups, with each comprised of 5-10 individuals. An additional 20 adolescents, 16-17 years of age who may or may not be sexually active (not asked for minors to disclose when screening) will be invited to participate in two focus groups designed to understand and compare perceptions and contraception decision making and choice of younger vs. older adolescents and young adults, anticipating differences in perception and behavior borne out in studies of AYA LARC uptake and contraceptive choice. A subsample of 22 focus group participants (18-21 years of age) will be invited to participate in an in-depth, individual interview designed to explore more intimate experiences and considerations related to relationships, feelings about their reproductive futures, personal issues related to living with their condition, and how culture and family influence their perceptions and use of contraception options.

In the interest of ensuring representation of young women living with a variety of chronic conditions, both visible and invisible, investigators will recruit AYA patients receiving care from the following subspecialty services:

* rheumatology (e.g., lupus, JIA, scleroderma, etc.)
* hematology (sickle cell disease, thalassemia)
* oncology (survivors)
* cardiology (congenital and acquired cardiac disease, including transplant)
* endocrinology (Type 1/2 diabetes)
* neurology (epilepsy, multiple sclerosis, cerebral palsy)
* pulmonology (cystic fibrosis)
* gastroenterology (inflammatory bowel disease, liver transplant)
* nephrology (chronic kidney disease, kidney transplant) and
* spina bifida

Focus groups with young adult women or transmale identified (have the potential for pregnancy) 18-21 years of age will be organized into groups of patients sharing the same condition (e.g., sickle cell disease, cystic fibrosis, etc.) or receiving care from the same subspecialty service, (e.g., pulmonology, nephrology, etc.). The groups will also be organized by sexually active and non-sexually active if there are a large number of adult aged participants who have not engaged in sexual activity. The team will randomly select two patients per subspecialty to be invited to participate in individual in-depth interviews.

The two focus groups with younger adolescent patients 16-17 years of age will include representation from each of the targeted subspecialty services (i.e. a mix of medical conditions), approximately two patients per subspecialty.

Findings from this study will inform the development of improved and more patient-centered counseling that takes into account these numerous intersecting factors. It will also contribute to the development of improved continuing education for pediatric specialty providers around the sexual and reproductive health needs of their patients, grounded in a cultural humility model and reproductive justice framework. Investigators expect that these, in turn, will contribute to better and more just sexual and reproductive health outcomes for medically complex AYA.

ELIGIBILITY:
Inclusion Criteria:

* 16-21 years of age
* female or transmale identified (i.e. have potential for pregnancy)
* ICD9/10 diagnostic codes corresponding with chronic illness/disability from the following CHLA subspecialty services:
* rheumatology (e.g., lupus, JIA, scleroderma, etc.)
* hematology (sickle cell disease, thalassemia)
* oncology (survivors)
* cardiology (congenital and acquired cardiac disease, including transplant)
* endocrinology (Type 1/2 diabetes)
* neurology (epilepsy, multiple sclerosis, cerebral palsy)
* pulmonology (cystic fibrosis)
* gastroenterology (inflammatory bowel disease, liver transplant)
* nephrology (chronic kidney disease, kidney transplant) and
* spina bifida multidisciplinary clinic
* Receiving ongoing care (at least one visit per year for more than one year) in one of the ten sub-specialty services targeted for the study
* English speaking
* Cognitive capacity for participation in a group discussion with other AYA, or an individual interview, about contraception
* Access to a phone, tablet or computer that has camera/video capabilities and willing to download the video conference platform in order to participate in the study procedures

Parent/caregiver Inclusion Criteria (parents/caregivers of minor participants)

* Legal parent/caregiver of patient 16-17 years old meeting study criteria
* English or Spanish speaking

Exclusion Criteria:

* Patients from the above sub-specialty services less than 16 years of age or greater than 21 years of age
* Non-English speaking
* Consult patients or patients who have not received ongoing care (i.e., care at least one visit per year for more than one year) from these subspecialty services
* Neurocognitive disability
* Patients with known infertility and/or history of receiving gonadotoxic therapies, for whom childbearing is known to be impossible
* Patients who do not have access to digital platforms necessary to participate in the study

Parent/caregiver Exclusion Criteria (parents/caregivers of minor participants)

* Adult accompanying patient who is not legal parent/caregiver
* Non-English/non-Spanish speaking

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent and young adults with a chronic condition being treated at Children's Hospital Los Angeles
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
This research will identify chronically ill individuals experiences with sexual and reproductive health patient-centered counseling from their subspecialty providers | Immediately after the focus groups and analysis have been completed
  Findings from this study will inform the development of improved and more patient-centered counseling that takes into account the numerous intersecting factors CHLA patients experience. By hearing first-hand experiences from patients, investigators will be able to identify the gaps in knowledge and care as it pertains to the sexual and reproductive health of patients with chronic medical conditions.
Focus groups will help identify gaps and areas for continuing education for pediatric sub-specialty providers as it pertains to the sexual and reproductive health of their patients | Immediately after the focus groups and analysis have been completed
  This research will contribute to the development of improved continuing education for pediatric specialty providers around the sexual and reproductive health needs of their patients, grounded in a cultural humility model and reproductive justice framework. By hearing from patients' experiences, investigators will be able to identify the areas that providers require extra knowledge or support to better educate their patients about their own sexual and reproductive health, especially as it relates to their chronic condition.

SECONDARY OUTCOMES:
This research will identify how to improve sexual and reproductive health outcomes for medically complex AYAs | Immediately after the focus groups and analysis have been completed
  This research will contribute to better and more just sexual and reproductive health outcomes for medically complex adolescent and young adults by providing first-hand patient experience to learn and improve from.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Borzutzky, MD, Principal Investigator — Children's Hospital Los Angeles; Ellen Iverson, MPH, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers